CLINICAL TRIAL: NCT00179764
Title: Immunoablative Protocol for Allogeneic Related and Unrelated Hematopoietic Peripheral Blood Stem Cell Transplant (HPBSC)
Brief Title: Immunoablative Mini Transplant (Hematopoietic Peripheral Blood Stem Cell Transplant [HPBSC])
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Reggie E Duerst, MD, MD, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT 0300 Mini
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Tumors; Malignant Melanoma; Hematological Malignancies; Myelogenous Leukemia, Chronic; Leukemia, Lymphoblastic, Acute
Keywords: Patients with recurrent solid tumors; Patients with malignant melanoma; Patients with hematological malignancies; Acute lymphoblastic leukemia (ALL); Acute myelogenous leukemia (AML)
MeSH Terms: conditions — Neoplasms; Melanoma; Hematologic Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Nurse Clinicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reduced Intensity Conditioning Regimen (Other)
  Interventions: Procedure: Immunoablative Hematopoietic PBSC Transplant; Procedure: Busulfan pharmacokinetics; Radiation: Central Nervous System (CNS) prophylaxis radiation

INTERVENTIONS:
Procedure: Immunoablative Hematopoietic PBSC Transplant — Immunoablative conditioning chemotherapy regimen, followed by transplantation of peripheral blood stem cells on Day 0 of the conditioning regimen.
Procedure: Busulfan pharmacokinetics — Pharmacokinetics of once-a-day dosing of intravenous busulfan as a 3-hour infusion
Radiation: Central Nervous System (CNS) prophylaxis radiation — * Patients diagnosed with ALL over 1 year of age and without prior CNS disease will receive CNS prophylaxis radiation to the whole brain prior to transplant.
  * Patients diagnosed with ALL with prior CNS disease over the age of 1 year will be treated with prophylaxis radiation to the whole brain and spine prior to transplant.

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of transplantation of high doses of peripheral blood stem cells (stem cells are special cells found in the blood and bone marrow that produce new blood cells) after treatment with non-myeloablative chemotherapy (not toxic to the bone marrow). In addition, this study will assess the side effects of the transplant.

DETAILED DESCRIPTION:
The standard treatment in many disorders of the bone marrow is high dose chemotherapy and whole-body radiation treatment followed by the stem cell transplant. This type of transplant not only suppresses or kills off the immune system, but is very toxic to the bone marrow. This study uses a chemotherapy regimen that will suppress the patient's immune system; however, it is non-myeloablative (not toxic to the bone marrow). It does not use whole-body radiation treatment. This approach can minimize the short- and long-term effects of transplantation. Other studies have shown that using chemotherapy followed by bone marrow transplantation without whole-body radiation can produce similar results as treatment with whole-body radiation.

Patients will be given chemotherapy with Fludarabine and Busulfan prior to the stem cell transplant. This treatment not only destroys diseased cells, but it also kills normal bone marrow cells. Following this experimental treatment, the patient will be given the stem cells through a central venous catheter (tube inserted in a vein). When the healthy stem cells are given to the patient, they will replace the destroyed bone marrow cells and produce new blood cells. The Allogeneic (not one's own) stem cells used in this experimental transplant will be obtained from a related matched donor or from an unrelated matched donor located through the National Marrow Donor Program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent solid tumors
* Patients with malignant melanoma
* Patients with hematological malignancies.

  * Chronic myelogenous leukemia in chronic or accelerated phase, to include chronic myelomonocytic leukemia (juvenile chronic myelogenous leukemia (JCML) or CMML).
  * Acute lymphoblastic leukemia (ALL)

    * First remission high-risk ALL (Ph+ with initial high white blood cell (WBC)t (4-11) in infants less than 1 year and CALLA negative)
    * Second or subsequent remission ALL or isolated extramedullary disease on or off therapy.
  * Acute non-lymphocytic leukemia (ANLL)

    * Patients with ANLL in first remission who have a matched sibling donor.
    * ANLL in second remission, or patients who only achieve an initial partial remission < 15% blasts, or early relapse.
  * Myelodysplastic syndromes (MDS): refractory anemia (RA), refractory anemia with excess blasts (RAEB), refractory anemia with excess blasts in transformation (RAEB-T) and CMML/JCML.
* Selected immunodeficiencies:

  * Wiskott-Aldrich syndrome.
  * Severe combined immunodeficiency variants that require ablation.
  * Hyper-Immunoglobulin M (IgM) syndrome.
  * Other immune deficiencies after approval from the medical director.
* Bone marrow failure syndromes (single or multiple hematopoietic lines)
* Venous access: A double lumen central vascular access device or its equivalent will be required for all patients entered on the protocol.
* Informed consent: The donor and the patient and/or the patient's legally authorized guardian must acknowledge in writing that consent to become a study subject has been obtained in accordance with the institutional policy approved by the United States (U.S.) Department of Health and Human Services.
* Patient organ function requirements:

  * Adequate renal function: serum creatinine < 2 x normal, or creatinine clearance calculated by Schwartz formula, of glomerular filtration rate (GFR) > 40 ml/min/1.73m2, or an equivalent GFR as determined by the institutional normal range.
  * Adequate liver function: total bilirubin </= 2 x normal; and Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) </= 4 x normal.
  * Adequate cardiac function: shortening fraction of > 24% by echocardiogram, or ejection fraction of > 30% by radionuclide angiogram.
  * Adequate pulmonary function: Diffusion Lung Capacity Carbon Monoxide (DLCO), Forced Expiratory Volume in 1 second (FEV1) / Forced Vital Capacity (FVC) > 30% by pulmonary function test. For children who are uncooperative for pulmonary function tests and have no evidence of dyspnea at rest or exercise intolerance, pulse oximetry > 94% on room air is considered acceptable.
  * Performance status: Lansky Score >/= 60% for children </= 16 years of age; or Karnofsky > 60% status for those > 16 years of age.

Exclusion Criteria:

* Patients who are pregnant
* Inability to find a suitable donor for the patient
* Patient is HIV-positive
* Patient has active Hepatitis B
* Disease progression or relapse prior to HPC infusion

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2000-03-10 (Actual); Primary Completion 2014-01-24 (Actual); Study Completion 2014-01-24 (Actual)

PRIMARY OUTCOMES:
Evaluate the morbidity and mortality of matched related and unrelated hematopoietic progenitor cell (HPC) transplantation at Children's Memorial Hospital using high dose CD34+ HPCs after a reduced intensity conditioning regimen. | To study end
Determine the toxicity of a reduced intensity conditioning regimen consisting of Fludarabine and Busulfan. | To study end

SECONDARY OUTCOMES:
Validate the pharmacokinetics of once-a-day dosing of intravenous Busulfan given as a 3-hour infusion, using a limited number of samples. | To study end
Assess chimeric engraftment utilizing this regimen in malignant and non-malignant disorders. | To study end
Assess the relapse rate of patients transplanted with this reduced intensity regimen. | To study end
Determine the incidence of acute and chronic Graft vs. Host Disease (GVHD) using prophylaxis with Cyclosporine A and mycophenolate mofetil following this reduced intensity regimen. | To study end

CONTACTS AND LOCATIONS:
Overall Officials: Morris Kletzel, M.D., Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Lurie Children's Hospital, Chicago, Illinois, United States